CLINICAL TRIAL: NCT03244917
Title: Trial to Reduce Antimicrobial Use In Nursing Home Residents With Alzheimer's Disease and Other Dementias (TRAIN-AD)
Brief Title: Trial to Reduce Antimicrobial Use In Nursing Home Residents With Alzheimer's Disease and Other Dementias
Acronym: TRAIN-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Susan Mitchell, MD, Senior Scientist, Hebrew SeniorLife
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: TRAIN-AD
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Dementia; Infection, Bacterial
Keywords: Nursing home; Palliative Care; Dementia; Infection; Antimicrobials
MeSH Terms: conditions — Dementia; Bacterial Infections; Infections

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research assistants collecting outcome data through chart reviews and follow-up proxy interviews will be blinded to nursing home randomization. The Principal Investigator, data programmers, and statistician will be blinded to treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRAIN-AD (Experimental): The study intervention is a multi-component training and education program targeting direct care providers and healthcare proxies for advanced dementia NH residents, intended to improve the management of urinary and lower respiratory tract infections in advanced dementia patients. There are two components to this practice intervention: 1. Provider Training, and 2. Proxy Education.
  Interventions: Behavioral: TRAIN-AD
- CONTROL (No Intervention): Facility randomized to the control arm will employ usual care for the management for suspected infections in advanced dementia,

INTERVENTIONS:
Behavioral: TRAIN-AD — The study intervention is a multi-component training and education program targeting direct care providers and healthcare proxies for advanced dementia NH residents, intended to improve the management of urinary and lower respiratory tract infections in advanced dementia patients. There are two components to this practice intervention: 1. Provider Training, and 2. Proxy Education. Intervention components aimed at the provider include: Professionally led infection management training seminars, online infection management course, and infection management guidance algorithms. Additionally participating prescribing providers will be sent bimonthly infection management feedback reports. Proxy Education is completed by providing an infection management in Advanced Dementia booklet to proxies of patients with AD upon resident enrollment in study.
  Arms: TRAIN-AD

SUMMARY:
This is a 52-month study (8 months preparation; 36 months to conduct the trial; 8 months data analyses and manuscript preparation) of a cluster randomized controlled trial (RCT) of an intervention to improve infection management for suspected UTIs and LRIs among residents with advanced dementia (N=480; N=240/arm) living in NHs (N=24; N=12/arm). The NH is the unit of randomization as the intervention must be delivered at the facility level to avoid contamination and because this is how it would be employed in the real-world. Analyses will be at the patient level.

DETAILED DESCRIPTION:
The final stage of dementia is characterized by recurrent suspected infections. Research has shown these episodes are widely mismanaged, leading to adverse patient and public health outcomes. Antimicrobials are extensively prescribed in advanced dementia, most often in the absence of clinical evidence to support a bacterial infection. Antimicrobial exposure is the main risk factor for multidrug-resistant organisms (MDROs). Nursing home (NH) residents with advanced dementia are three times more likely to be colonized with MDROs compared to other residents. Moreover, as these patients are in the terminal phase of dementia, evidence suggests they may not clinically benefit from antimicrobials. Comfort is the stated goal of care for 90% of advanced dementia patients, and the risks and burdens associated with work-up and treatment of suspected infections generally do not promote that goal, particularly when hospitalization is involved. Taken together, there is a clear need to improve infection management in advanced dementia both to provide better end-of-life care to these patients and reduce the public health threat of MDROs.

This is a 52-month study (8 months preparation; 36 months to conduct the trial; 8 months data analyses and manuscript preparation) of a cluster randomized controlled trial (RCT) of an intervention to improve infection management for suspected UTIs and LRIs among residents with advanced dementia (N=410; N=205/arm) living in NHs (N=28; N=14/arm). The NH is the unit of randomization as the intervention must be delivered at the facility level to avoid contamination and because this is how it would be employed in the real-world. Analyses will be at the patient level.

ELIGIBILITY:
Inclusion Criteria:

Facility inclusion criteria

1. More than 60 beds
2. Within 60 miles of Boston

Resident inclusion eligibility criteria

* Age > or = to 60 years
* A diagnosis of dementia (any type)
* Global Deterioration Scale (GDS) score of 7
* NH length of stay >90 days
* An individual who can communicate in English has been formally or informally designated as a health care proxy
* Not comatose GDS stage 7 features include: profound memory deficits (cannot recognize family), total functional dependence, speech <= 5 words, incontinence, and non-ambulatory. GDS 7 was chosen to define advanced dementia as it has been successfully operationalized and validated in or prior studies, and experts agreed to use this definition in research studies. A 90 day minimum length of stay was chosen to exclude short-stay patients.

Provider inclusion criteria

* Direct care provider of advanced dementia residents (a nurse, nurse practitioner, physician or physician assistant identified by a senior administrator as an individual who cares for residents with advanced dementia)
* Can communicate in English (because intervention materials are all in English),
* Over 21 years of age.

Exclusion Criteria:

Residents with cognitive impairment due to causes other than dementia (e.g., head trauma and in short-term, sub-acute SNFs) will be excluded.

Residents' whose proxies cannot communicate in English will be excluded from the study, because the information directed to proxies are only in English.

Providers that do not provide direct care to residents with advanced dementia or who do not speak English.

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Mitchell, MD. MPH, Principal Investigator — Hebrew SeniorLife
Locations (1):
- Hebrew SeniorLife, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitchell SL, D'Agata EMC, Hanson LC, Loizeau AJ, Habtemariam DA, Tsai T, Anderson RA, Shaffer ML. The Trial to Reduce Antimicrobial Use in Nursing Home Residents With Alzheimer Disease and Other Dementias (TRAIN-AD): A Cluster Randomized Clinical Trial. JAMA Intern Med. 2021 Sep 1;181(9):1174-1182. doi: 10.1001/jamainternmed.2021.3098. PMID 34251396
- [Derived] Shaffer ML, D'Agata EMC, Habtemariam D, Mitchell SL. Covariate-constrained randomization for cluster randomized trials in the long-term care setting: Application to the TRAIN-AD trial. Contemp Clin Trials Commun. 2020 Mar 17;18:100558. doi: 10.1016/j.conctc.2020.100558. eCollection 2020 Jun. PMID 32258819
- [Derived] Loizeau AJ, D'Agata EMC, Shaffer ML, Hanson LC, Anderson RA, Tsai T, Habtemariam DA, Bergman EH, Carroll RP, Cohen SM, Scott EME, Stevens E, Whyman JD, Bennert EH, Mitchell SL. The trial to reduce antimicrobial use in nursing home residents with Alzheimer's disease and other dementias: study protocol for a cluster randomized controlled trial. Trials. 2019 Oct 15;20(1):594. doi: 10.1186/s13063-019-3675-y. PMID 31615540

RESULTS

PARTICIPANT FLOW:
Groups:
- TRAIN-AD: Residents with advanced dementia living in nursing homes randomized to receive the TRAIN-AD program to guide the management of suspected urinary and respiratory tract infections
- Control: Residents with advanced dementia living in facilities randomized to control arm that employed usual care to manage suspected urinary and respiratory tract infections
Period: Overall Study
Arm/Group | TRAIN-AD | Control
Started | 201 | 229
Completed | 199 | 227
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRAIN-AD | Control | Total
Number analyzed (Participants) | 199 | 227 | 426
Age, Continuous [Mean (Standard Deviation); unit: years] | 87.7 (8.0) | 85.3 (8.6) | 86.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 190 | 353
  Male | 36 | 37 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 22 | 49
  White | 166 | 200 | 366
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Total Antimicrobial Use for LRI and UTIs
Description: The investigators will compare the total number of antimicrobial courses for suspected UTIs and LRIs/person-year (primary outcome) over 12 months in the intervention vs. control (usual care) arms. Data will be obtained from review of the residents' charts and medication administration records q2months up to 12 months
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: antimicrobial courses per person-year
Arm/Group | TRAIN-AD | Control
Number analyzed (Participants) | 199 | 227
antimicrobial courses per person-year | 0.55 [0.25 to 0.84] | 0.82 [0.49 to 1.14]

2. Secondary Outcome: Antimicrobial Use When Minimal Criteria Are Absent for LRI and UTIs
Description: The investigators will compare the number of antimicrobial courses prescribed for suspected UTIs and LRIs when minimal criteria for treatment initiation are absent based on consensus guidelines/person-year (secondary outcome) in the intervention vs. control arm over 12 months.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: antimicrobial courses per person-year
Arm/Group | TRAIN-AD | Control
Number analyzed (Participants) | 199 | 227
antimicrobial courses per person-year | 0.37 [0.15 to 0.60] | 0.43 [0.23 to 0.62]

3. Secondary Outcome: Burdensome Interventions
Description: The investigators will compare the number of burdensome procedures used to evaluate suspected LRIs and UTIs (hospital transfer, bladder catheterization, chest x-ray, blood draws)/person-year between the intervention versus control arm
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: interventions per person-year
Arm/Group | TRAIN-AD | Control
Number analyzed (Participants) | 199 | 227
interventions per person-year | 1.07 [0.54 to 1.60] | 1.69 [0.87 to 2.51]

4. Secondary Outcome: Total Antimicrobial Use
Description: The investigators will compare the total number of antimicrobial courses prescribed for any reason /person-year over 12 months in the intervention vs. control (usual care) arms. Data will be obtained from review of the residents' charts and medication administration records q2months up to 12 months
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: antimicrobial courses per person-year
Arm/Group | TRAIN-AD | Control
Number analyzed (Participants) | 199 | 227
antimicrobial courses per person-year | 0.82 [0.52 to 1.13] | 1.19 [0.83 to 1.56]

ADVERSE EVENTS:
Time Frame: Each residents was followed for up to one year
Description: There were no pre-specified adverse events in this minimal risk study
Arm/Group | TRAIN-AD | Control
All-Cause Mortality (participants affected / at risk) | 82/199 | 102/227
Serious Adverse Events (participants affected / at risk) | 0/199 | 0/227
Other Adverse Events (participants affected / at risk) | 0/199 | 0/227

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT03244917/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03244917/SAP_001.pdf